CLINICAL TRIAL: NCT03094507
Title: The Pharmacokinetics of Dolutegravir, Darunavir/Cobocistat When Co-administered in Healthy Volunteers
Acronym: SSAT073
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St Stephens Aids Trust (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SSAT073
Record Dates: First submitted 2017-03-03; First posted 2017-03-29 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: HIV
MeSH Terms: interventions — dolutegravir; cobicistat mixture with darunavir

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group One (Experimental): Tivicay (Dolutegravir 50 mg) for 14 days OD (days 1-14) WASH OUT for 7 days (days 15-21) Tivicay (Dolutegravir 50 mg) OD plus Rezolsta (darunavir/cobicistat 800/150 mg) OD for 14 days (days 22-35) WASH OUT for 7 days (days 36-42) Rezolsta (darunavir/cobicistat 800/150 mg) OD for 14 days (days 43-56)
  Interventions: Drug: Tivicay; Drug: Rezolsta
- Group Two (Experimental): Rezolsta (darunavir/cobicistat 800/150 mg) OD for 14 days (days 1-14) WASH OUT for 7 days (days 15-21) Tivicay (Dolutegravir 50 mg) OD plus Rezolsta (darunavir/cobicistat 800/150 mg) OD for 14 days (days 22-35) WASH OUT for 7 days (days 36-42) Tivicay (Dolutegravir 50 mg) for 14 days OD (days 43-56)
  Interventions: Drug: Tivicay; Drug: Rezolsta

INTERVENTIONS:
Drug: Tivicay — 50 mg once daily
  Other Names: Dolutegravir
Drug: Rezolsta — darunavir 800 mg/cobicistat 150 mg once daily
  Other Names: darunavir/cobicistat

SUMMARY:
The purpose of this study is to look at the levels of three HIV medications: dolutegravir, darunavir and cobicistat in the blood after drug intake has been stopped, in order to understand how long these drugs persist in the blood. The study will specifically look at blood levels of these three drugs after taking them every day for 14 days.

There will be two groups. Participants in Group 1 will take dolutegravir everyday for 14 days, then nothing for 7 days, then dolutegravir and darunavir/cobicistat together for 14 days, nothing for 7 days, and then darunavir/cobicistat alone for 14 days. If participants go into Group 2 they will begin with darunavir/cobicistat everyday for 14 days, then nothing for 7 days, then dolutegravir and darunavir/cobicistat together for 14 days, nothing for 7 days, and then dolutegravir alone for 14 days. Drug levels for both groups will be measured on days 14, 35 and 56. If the participants decide to take part, the duration of the study will be up to 57 days plus a screening visit which will take place up to 28 days prior to the start of the study, and a follow up visit, which takes place 15 to 22 days after the last dose of study medication. Eligible participants will be randomized (1:1 ratio) to group 1 or group 2. Participants and the study doctor will know which study medications the participant is taking at all times during the study.

DETAILED DESCRIPTION:
This is a randomised, cross-over, open label study, which means that the participants will be randomly assigned to the different arms of the study which receive different medications. The participants and the study doctor will know which study medications the participant is taking at all times during the study.This study will be conducted in a single site, in London.

The total duration of the participant's involvement in the study will be up to 57 days plus a screening visit up to 28 days prior to the start of the study, and a follow up visit 27 to 33 days after the last blood measurement.

The participants will be asked to visit the clinic on up to 14 occasions, of which three visits involve staying in the unit for approximately 12 hours (day 14,35 and 56).

Blood samples will be taken from the participants throughout the study to measure the levels of dolutegravir, darunavir and cobicistat in blood. Blood and urine will also be collected throughout the study for safety analysis; this is to ensure the participants are healthy to take part or to continue taking part in the study. The total amount of blood collected from each participant during the study will be approximately 500ml (just below a pint).

Participants will be provided with written information about the study in the form of a participant information sheet and will be allowed adequate time for questions and to consider the study before agreeing to participate. It will be the responsibility of the investigator or the co-investigator to obtain written informed consent prior to undertaking any procedure detailed in the protocol. As part of the consent procedure, participants will also be asked consent to their personal details being entered into TOPS (the over-volunteering protection system).

The investigator or designee will provide adequate explanation of the aims, methods, objectives and potential hazards of the study. They will also be explaining to the participants that they are free to refuse or withdraw from the study for any reason without detriment to their future care or treatment.

A detailed description of each study visit follows below:

1. Screening visit If the participant agrees to take part, they will firstly be asked to sign the informed consent form and they will be given a copy to keep.

   During the visit the following assessments will be carried out:

   • Demographic details

   • Full medical, drug and social history

   • Physical examination including weight, height, and vital signs (temperature, blood pressure, heart rate, and respiratory rate)

   • ECG

   • Chemistry panel

   • Haematology with a differential and clotting screen

   • HIV antibody testing

   • Hepatitis B and C screening

   • Urinalysis (macro analysis)

   • Drug screen (urine)

   • Pregnancy test (urine) for WOCBP (women of child-bearing potential)

   • Registration of TOPS database

   • Concomitant medications

   GP verification of medical history: A medical history questionnaire will be sent to all participants' GPs for verification of medical history. This information will be reviewed by the Investigator as part of the medical history evaluation. If the completed questionnaire is not received from the GP, then the available information regarding the participant will be reviewed by the Investigator. The Investigator will assess this information and decide whether they are sufficiently confident that the inclusion and exclusion criteria are met and whether the participant may be enrolled into the study. This decision must be documented in writing BEFORE the participant is dosed. Copies of sent GP letters and returned confirmation of medical history will be filed in each participant's source documentation.
2. Baseline Visit, Day 1

   Participants will attend the Unit in the morning and will be asked to fast for 8 hours overnight prior to attending. The following evaluations will be performed in the morning of Day 1, before study medication dosing:

   • Vital signs (temperature, blood pressure, heart rate, and respiratory rate)

   • Haematology with a differential and clotting screen

   • Chemistry panel

   • Urinalysis (macro analysis)

   • Pregnancy test for WOCBP (urine)

   • Drug screen (urine)

   • Concomitant medications

   • Review of adverse events (AEs) Blood samples will be collected for:

   - Laboratory tests for safety

   - Pharmacogenetics if they have agreed to this part of the study

   - Platelets function (to investigate how clotting works in people taking anti-HIV medication).

   Group1:

   A Tivicay® (dolutegravir) tablet will be administered with a standard breakfast, made up according to instructions along with 240 ml of water. This will set the nominal time of dosing. Subjects will be instructed to administer Tivicay® at home in the morning on all other days (14 days in total) (with the exception of days 7, and 14, when the drug will be administered in the PK Unit). Participants will be instructed to administer study drugs in the morning within 15 min of standard breakfast.Participants will be given a diet sheet giving examples of a standardised breakfast for them to have at home with the study drug. They will be also reminded to take their study drug to the unit on day 14 as they will take their last dose in the unit on that day.

   Group2:

   A Rezolsta® (darunavir plus cobicistat) tablet will be administered with a standard breakfast, made up according to instructions along with 240 ml of water. This will set the nominal time of dosing. Subjects will be instructed to administer Rezolsta® at home in the morning on all other days (14 days in total) (with the exception of days 7, and 14, when the drug will be administered in the PK Unit). Subjects will be instructed to administer study drugs in the morning within 15 min of standard breakfast.Participants will be given a diet sheet giving examples of a standardised breakfast for them to have at home with the study drug. They will be also reminded to take their study drug to the unit on day 14 as they will take their last dose in the unit on that day.
3. Wash out periods (Days 15 to 21 and Days 36 to 42):Group 1 and 2

From days 15 to 21 and days 36 to 42, participants will be asked to stop taking their study medication for a total of 7 days each time. These are the washout periods. 7) Intensive Pharmacokinetic Visits (Days 14, 35 and 56) Participants will be admitted to the unit in the morning on days 14, 35 and 56 and will remain in the Unit for approximately 12 hours. They will be asked to fast for 8 hours overnight prior to attending.

The following evaluations will be performed in the morning of Days 14, 35 and 56, before study medication dosing: Vital signs (temperature, blood pressure, heart rate, and respiratory rate) • Physical Examination (symptom directed)

• Adherence questioning

* Review of AEs
* Concomitant medication check
* Haematology with a differential and clotting screen
* Chemistry panel
* Urinalysis (macro analysis)
* Drug screen (urine)
* Pregnancy test for WOCBP (urine)
* Pill count
* Blood samples will be collected for:Platelets function (to investigate how clotting works in people taking anti-HIV medication).

Serial blood samples will be taken on 6 occasions over the day (pre-dose (within 10 minutes before dosing), then 2, 4, 6, 8, and 12 hrs later) to measure the levels of study drugs in their blood. A cannula will be placed in a vein in the participant's forearm to allow repeated blood samples to be taken without having to repeatedly use a needle.

The exact time of intake of study medication will be recorded on the CRF. Participants should remain in a semi- recumbent position until four hours post dose.

Patients will be able to leave the unit after the 12 hour sample to return the following morning.

• Tail Pharmacokinetic Visits (Day 15, 36 and 57)

Participants will be required to attend the unit for plasma drug concentration sampling. This will occur at 24 hours post dose.

Participants will attend on days 5, 36 and 57.

• Follow up visit (day 84 to 90)

Participants will return to the unit on one occasion between days 80 to 90 inclusive and undergo the following evaluations:

* Vital signs (temperature, blood pressure, heart rate, and respiratory rate)
* Haematology with a differential and clotting screen
* Chemistry panel.
* Concomitant medications
* Review of AEs

  10) Early termination visit In case of early termination, participants will attend the unit for an early termination visit within one week (or otherwise as the investigator believes appropriate).

During this visit the following evaluations will be performed:

* Vital signs (temperature, blood pressure, heart rate, and respiratory rate)
* Haematology with a differential and clotting screen
* Chemistry panel
* Concomitant medications and adverse event check The reason for the early termination of the participant will be clearly documented on the participant's CRF. The participant will not then be required to attend for a follow up visit unless deemed necessary in the opinion of the investigator (e.g. due to adverse event follow up).

ELIGIBILITY:
Inclusion Criteria:

1. The ability to understand and sign a written informed consent form, prior to participation in any screening procedures and must be willing to comply with all study requirements
2. Male or Non-pregnant, non-lactating females.
3. Between 18 to 65 years, inclusive
4. Body Mass Index (BMI) of 18 to 35 kg/m2, inclusive
5. ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). A single repeat is allowed for eligibility determination.
6. Women of childbearing potential (WOCBP - definition in Appendix 5) must be using an adequate method of contraception to avoid pregnancy throughout the study and for a period of at least 4 weeks after the study.

   A female may be eligible to enter and participate in the study if she:
   1. is of non-child-bearing potential defined as either post-menopausal (12 months of spontaneous amenorrhea and ≥ 45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy or,
   2. is of child-bearing potential with a negative pregnancy test at both Screening and Day 1 and agrees to use one of the following methods of contraception to avoid pregnancy:
   3. Complete abstinence from penile-vaginal intercourse from 2 weeks prior to administration of IP, throughout the study, and for at least 4 weeks after discontinuation of all study medications;
   4. Double barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide);
   5. Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year (not all IUDs meet this criterion, see protocol appendix 5 for an example listing of approved IUDs);
   6. Male partner sterilization confirmed prior to the female subject's entry into the study, and this male is the sole partner for that subject;
   7. Approved hormonal contraception (see protocol appendix 5 for a listing of examples of approved hormonal contraception) plus male condom;
   8. Any other method with published data showing that the expected failure rate is <1% per year.
   9. Any contraception method must be used consistently, in accordance with the approved product label and for at least 4 weeks after discontinuation of IP.
7. Men who have partners who are women of childbearing potential (WOCBP - definition in Appendix 5) must be using an adequate method of contraception to avoid pregnancy in their partner throughout the study and for a period of at least 4 weeks after the study (see inclusion criteria 6);

   * Complete abstinence from penile-vaginal intercourse
   * Double barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide);
   * Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year (not all IUDs meet this criterion, see Appendix 5 for an example listing of approved IUDs);
   * Male partner sterilization confirmed prior to the female subject's entry into the study, and this male is the sole partner for that subject;
   * Any other method with published data showing that the expected failure rate is <1% per year. and not containing hormones.

   Any contraception method must be used consistently, in accordance with the approved product label and for at least four weeks after discontinuation of IMP.
8. Willing to consent to their personal details being entered onto the TOPS database
9. Willing to provide proof of identity by photographic ID at screen and any subsequent visit
10. Registered with a GP in the UK

Exclusion Criteria:

1. Any clinically significant acute or chronic medical illness
2. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations
3. Positive blood screen for hepatitis B surface antigen or C antibody
4. Positive blood screen for HIV-1 or 2 by antibody/antigen assay
5. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
6. History or presence of allergy to the study drugs and their components: darunavir, cobicistat, dolutegravir or excipients (sodium methyl parahydroxybenzoate, lactulose, Hypromellose Colloidal silicon dioxide, Silicified microcrystalline cellulose Crospovidone, Magnesium stearate, Polyvinyl alcohol- partially hydrolysed, Macrogol 3350,Titanium dioxide, Talc, Iron oxide red, Iron oxide black, Lactose monohydrate, Magnesium stearate, Gelatine Yellow iron oxide, Indigocarmin (E132), White ink, Shellac,Titanium dioxide (E171), Ammonium hydroxide, Propylene glycol , Simethicone, Hypromellose, Polyvinyl alcohol-partially hydrolysed, Macrogol 3350) Mannitol (E421) Microcrystalline cellulose Povidone K29/32, Sodium starch glycolate, Sodium stearyl fumarate, Polyvinyl alcohol-partially hydrolyzed, Titanium dioxide (E171), Macrogol Talc Iron oxide yellow (E172)
7. Current or recent (within three months) gastrointestinal disease
8. Known intolerance of lactose monohydrate, sunset yellow aluminium lake (E110), and patients with galactose intolerance, the Lapp lactase deficiency, or glucose-galactose malabsorption
9. Clinically relevant alcohol or drug use (positive urine drug screen) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance with treatment, follow-up procedures or evaluation of adverse events. Smoking is permitted, but tobacco intake should remain consistent throughout the study
10. Exposure to any investigational drug (or placebo) or participation in a clinical study involving the donation of blood samples within three months of first dose of study drug
11. Use of any other drugs (unless approved by the Investigator), including over-the-counter medications and herbal preparations, within two weeks prior to first dose of study drug, unless approved/prescribed by the Principal Investigator as known not to interact with study drugs.
12. Females of childbearing potential without the use of effective non-hormonal birth control
13. Methods, or not willing to continue practising these birth control methods for at least four weeks after the end of the treatment period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2018-01-17 (Actual); Study Completion 2018-03-17 (Actual)

PRIMARY OUTCOMES:
Assess the pharmacokinetics of dolutegravir and darunavir/cobicistat during co-administration in HIV negative healthy volunteers as measured by Cthrough | 8 weeks
  Trough concentration (Ctrough) is defined as the concentration at 24 hours after the observed drug dose
Assess the pharmacokinetics of dolutegravir and darunavir/cobicistat during co-administration in HIV negative healthy volunteers as measured by Cmax | 8 weeks
  Cmax defined as the maximum observed plasma concentration.
Assess the pharmacokinetics of dolutegravir and darunavir/cobicistat during co-administration in HIV negative healthy volunteers as measured by t1/2 | 8 weeks
  t1/2 = Elimination half-life
Assess the pharmacokinetics of dolutegravir and darunavir/cobicistat during co-administration in HIV negative healthy volunteers as measured by Tmax | 8 weeks
  Tmax = time point at Cmax
Assess the pharmacokinetics of dolutegravir and darunavir/cobicistat during co-administration in HIV negative healthy volunteers as measured by total drug exposure | 8 weeks
  Total drug exposure is expressed as the area under the plasma concentration-time curve from 0-24 hours after dosing (AUC0-24h)

SECONDARY OUTCOMES:
Assess the safety and tolerability of the studied drugs when co-administered to HIV negative healthy volunteers, assessed by The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events | 10 weeks
  studied drug: Dolutegravir and Darunavir/Cobocistat
investigate the association between genetic polymorphisms in drug disposition genes and drug exposure as measured by Peak plasma concentration (Cmax) | 8 weeks
  investigate the association between genetic polymorphisms in drug disposition genes and drug exposure
investigate the association between genetic polymorphisms in drug disposition genes and drug exposure as measured by trough concentration (Ctrough) | 8 weeks
  investigate the association between genetic polymorphisms in drug disposition genes and drug exposure
investigate the association between genetic polymorphisms in drug disposition genes and drug exposure as measured by Area under the plasma concentration versus time curve (AUC) | 8 Weeks
  investigate the association between genetic polymorphisms in drug disposition genes and drug exposure
Exploratory: the impact of antiretroviral drugs on platelet function | 8 weeks
  To look at platelet function during antiretroviral intake in HIV negative individuals who take part in clinical trials. Platelet aggregation response as a change in light transmission in a platelet aggregometer, will be measured. The data reported will be the maximal aggregation in response to agonist stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, Principal Investigator — St Stephen's AIDS Trust
Locations (1):
- St Stephen's Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Only authorised representatives of the sponsor (such as monitors and auditors) and individuals who are authorised on the signature and delegation log will have access to the participants' personal data. This could typically be: doctors, nurses, pharmacists, laboratory staff and data manager within the Trust/Care organisation. It is also possible that the regulatory authorities may wish to access this data. The access given to participants' data is explained in the participant information sheet, so consent will have been given to these individuals outside the care organisation.